CLINICAL TRIAL: NCT05267626
Title: A Phase 1/2, First-in-Human, Open Label, Dose Escalation and Expansion Study of AU-007, A Monoclonal Antibody That Binds to IL-2 and Inhibits IL-2Rα Binding, in Patients With Unresectable Locally Advanced or Metastatic Cancer
Brief Title: Study of AU-007, A Monoclonal Antibody That Binds to IL-2 and Inhibits IL-2Rα Binding, in Patients With Unresectable Locally Advanced or Metastatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aulos Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-AU-007-01
Record Dates: First submitted 2022-02-10; First posted 2022-03-04 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor; Metastatic Cancer; Cutaneous Melanoma; Non-Small Cell Lung Cancer
Keywords: IL-2 CD25; IL-2Ra; Melanoma; Head and neck squamous cell carcinoma; Urothelial cancer; Gastric Cancer; Gastro-esophageal cancer; CD25; IL-2; NSCLC; Bladder Cancer; Merkel Cell Cancer; Proleukin; Immune Therapy; Immunotherapy; Cutaneous Squamous Cell Cancer; Cytokine; Anti-PD-L1; Non-small cell lung cancer; Clear cell renal cell cancer
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma; Carcinoma, Non-Small-Cell Lung; Diabetes Mellitus, Insulin-Dependent, 10; Squamous Cell Carcinoma of Head and Neck; Stomach Neoplasms; Urinary Bladder Neoplasms; Carcinoma, Merkel Cell; Carcinoma, Renal Cell | interventions — aldesleukin; avelumab; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- AU-007 Monotherapy (Experimental): AU-007 (Q2w) administered as a monotherapy sequential ascending doses with each Dose Escalation Cohort
  (Complete; no longer enrolling)
  Interventions: Drug: AU-007
- AU-007 combined with a single dose of aldesleukin (Experimental): AU-007 (Q2w) administered in combination with a single dose of aldesleukin with the initial AU-007 dose.
  Interventions: Drug: AU-007; Drug: Aldesleukin
- AU-007 combined with aldesleukin given concomitantly (Experimental): AU-007 administered in combination with aldesleukin, both administered Q2w
  (Complete; no longer enrolling)
  Interventions: Drug: AU-007; Drug: Aldesleukin
- AU-007 plus aldesleukin in combination avelumab (Experimental): AU-007 and avelumab administered Q2w with a single dose of aldesleukin with the initial AU-007 dose
  Interventions: Drug: AU-007; Drug: Aldesleukin; Drug: Avelumab
- AU-007 plus aldesleukin in combination with nivolumab (Experimental): AU-007 (Q2w) administered in combination with a single dose of aldesleukin with the initial AU-007 dose.
  Nivolumab will be administered Q4w.
  Interventions: Drug: AU-007; Drug: Aldesleukin; Drug: Nivolumab

INTERVENTIONS:
Drug: AU-007 — Monoclonal Antibody Targeting IL-2
Drug: Aldesleukin — IL-2
  Arms: AU-007 combined with a single dose of aldesleukin; AU-007 combined with aldesleukin given concomitantly; AU-007 plus aldesleukin in combination avelumab; AU-007 plus aldesleukin in combination with nivolumab
Drug: Avelumab — Monoclonal Antibody Targeting PD-L1
  Arms: AU-007 plus aldesleukin in combination avelumab
Drug: Nivolumab — Monoclonal Antibody Targeting PD-1
  Arms: AU-007 plus aldesleukin in combination with nivolumab

SUMMARY:
This is a first in human, open-label, multi-center Phase 1 / 2 study to evaluate the safety, tolerability, and initial efficacy of AU-007 in patients with advanced solid tumors. AU-007 will be administered either as a monotherapy, or in combination with a single loading dose of aldesleukin, or with both AU-007 and aldesleukin given every 2 weeks (Q2w). Once the recommended phase 2 dose (RP2D) of AU-007 plus aldesleukin was determined, (AU-007 Q2w plus a single loading dose of aldesleukin), AU-007 plus aldesleukin is also being administered with avelumab or nivolumab.

DETAILED DESCRIPTION:
This is a first in human, multicenter, open-label Phase 1-2 study evaluating the safety, tolerability, and initial efficacy of AU-007 with or without aldesleukin, in patients with unresectable locally advanced or metastatic cancer. Patients must either be ineligible for or have progressed on prior standard of care therapy.

Part 1 consists of 3 escalation Arms, each starting with a single 1+2 escalation cohort followed by 3+3 escalation cohorts to define the RP2D or maximum tolerated dose (MTD).

The study begins in Arm A evaluating escalating doses of AU-007 (Q2w) in sequential escalation cohorts to define RP2D or MTD.

In Arm B, AU-007 (Q2w) is evaluated in combination with a single dose of aldesleukin given with the first AU-007 dose. AU-007 is administered Q2w with an escalating single aldesleukin dose in sequential escalation cohorts.

In Arm C, AU-007 is evaluated in combination with aldesleukin, both given Q2w. AU-007 will be administered with an escalating dose of aldesleukin in each sequential Arm C escalation cohort.

The Part 2 cohort expansion portion of the study consists of up to three expansion Arms evaluating the initial efficacy of the RP2D (AU-007 plus a single loading dose of aldesleukin) in selected solid tumor types, prioritizing cutaneous melanoma and non-small cell lung cancer (NSCLC).

Part 3 evaluates the safety of AU-007 in combination with aldesleukin and avelumab, followed by one expansion cohort, in NSCLC.

Part 4 evaluates the safety of AU-007 plus aldesleukin in combination with nivolumab, followed by one expansion cohort, in cutaneous melanoma.

ELIGIBILITY:
Selected Inclusion Criteria:

* Patients must have measurable disease as per RECIST v1.1 criteria and documented by CT and/or MRI
* Part 2 includes but is not limited to:
* Cutaneous melanoma that is either locally unresectable or metastatic:

  * BRAF wild type: progressed after receiving PD-1 containing therapy with or without an anti-CTLA-4
  * BRAF mutation: patients who refused BRAF+MEK inhibitor
  * Must have objective progression after receiving at least two cycles of prior doublet therapy (anti-PD-1/anti-CTLA-4 or anti-PD-1/anti-LAG-3)
  * Radiographic progression ≥ 4 weeks prior to the first dose of study drug to rule out late response to most recent therapy. The requirement for documented radiologic progression may be waived after review by Medical Monitor (e.g., in the case of progression beyond 12 weeks after starting a doublet)
  * LDH ≤ 2.5 x ULN
* NSCLC: Unresectable locally advanced or metastatic PD-L1-positive (tumor proportion score [TPS] ≥ 1%) NSCLC not harboring an activating EGFR mutation or ALK rearrangement and has progressed during or following treatment with an anti-PDx with or without platinum-based chemotherapy
* Part 3: NSCLC as described above
* Part 4: cutaneous melanoma

  * Unresectable locally advanced or metastatic cutaneous melanoma that has progressed during or following treatment with an anti-PDx (unless ineligible for anti-PDx therapy)
  * Patients with BRAF mutations must either be ineligible for or have refused a BRAF+MEK inhibitor
  * Must have objective progression after receiving at least two cycles of prior doublet therapy (anti-PD-1/anti-CTLA-4 or anti-PD-1/anti-LAG-3).
  * Radiographic progression ≥ 4 weeks prior to the first dose of study drug to rule out late response to most recent therapy. The requirement for documented radiologic progression may be waived after review by Medical Monitor (e.g., in the case of progression beyond 12 weeks after starting a doublet)
  * LDH ≤ 2.5 x ULN
* Female patients of childbearing potential must have a negative serum or urine pregnancy test performed within 72 hours prior to the initiation of study drug administration. Female patients of childbearing potential must be willing to use two forms of contraception throughout the study, starting with Screening through 60 days after the last dose of study drug (or 5 months after the last dose of study drug for patients receiving nivolumab). Abstinence is acceptable if this is the established and the preferred contraception method for the patient
* Male patients with partners of childbearing potential must use barrier contraception from the time of consent through 60 days after discontinuation of study drug and must not donate sperm during this period. In addition, male patients should have their partners use contraception (as documented for female patients) for the same period of time
* Patients who have previously received an immune checkpoint inhibitor (e.g., anti-PD-L1, anti-PD-1, anti-CTLA-4) prior to enrollment must have checkpoint inhibitor immune-related toxicity resolved to either Grade ≤ 1 or baseline (prior to the checkpoint inhibitor) to be eligible for enrollment. Patients who experienced previous checkpoint inhibitor-related hypothyroidism are eligible for the study regardless of grade resolution if well controlled on thyroid hormone replacement therapy
* Symptomatic central nervous system (CNS) metastases must have been treated, be asymptomatic for ≥ 14 days, and meet the following at the time of enrollment:
* No concurrent treatment for CNS disease (e.g., surgery, radiation, corticosteroids ≥ 10 mg prednisone/day or equivalent)
* No concurrent leptomeningeal disease or cord compression

Exclusion Criteria:

* Patients with a history of known autoimmune disease with exceptions of

  * Vitiligo
  * Psoriasis, atopic dermatitis, or other autoimmune skin condition not requiring systemic treatment
  * History of Graves' disease in patients now euthyroid for > 4 weeks
  * Hypothyroidism managed by thyroid hormone replacement
  * Alopecia
  * Arthritis managed without systemic therapy beyond oral nonsteroidal anti- inflammatory drugs
* Major surgery or traumatic injury within 3 weeks before first dose of AU-007
* Unhealed wounds from surgery or injury
* Treatment with > 10 mg per day of prednisone (or equivalent) or other immune-suppressive drugs within the 7 days prior to the initiation of study drug. Steroids for topical, ophthalmic, inhaled, or nasal administration are allowed
* Prior anti-cancer therapy before the planned start of AU-007 as follows:

  * Not recovered to baseline from toxicity of prior systemic cancer therapy(ies).
  * Not recovered from toxicity of radiotherapy.
  * Concurrent use of hormones either to maintain castrate levels of testosterone in patients with castration-sensitive prostate cancer or for non-cancer-related conditions (e.g., insulin for diabetes, hormone replacement therapy) is acceptable. Bisphosphonates are permitted.
* Patients who have experienced serious adverse events during prior IL-2 therapy (including but not limited to bowel perforation, gastrointestinal bleeding, arrythmias, myocardial infarction, repetitive seizures).
* Inflammatory process that has not resolved for ≥ 4 weeks from the date of first study dose. Patients with chronic low-grade inflammatory processes such as radiation-induced pneumonitis are excluded regardless of duration
* Second primary invasive malignancy not in remission for ≥ 1 year. Exceptions include non-melanoma locally advanced skin cancer, cervical carcinoma in situ, localized prostate cancer (Gleason score ≤ 7), resected melanoma in situ, or any malignancy considered to be indolent and never required therapy, with the exception of indolent lymphomas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of AU-007 | Day 1 thru end of treatment (EOT) visit (28 days after last dose)
  Measured by the frequency of DLTs (Dose limiting toxicity) and safety profile
Establish the maximum tolerated dose (MTD) and/or RP2D | Day 1 thru EOT visit (28 days after last dose)
  With AU-007 alone or in combination with aldesleukin measured by pharmacokinetics (PK), pharmacodynamics (PD), and Biomarkers

SECONDARY OUTCOMES:
Magnitude of PK changes in the blood after dosing determined by area under the curve (AUC) of AU-007 | Day 1 thru EOT visit (28 days after last dose)
  The AUC of AU-007 will be measured at different timepoints after AU-007 administration
Magnitude of PK changes in the blood after dosing determined by maximum concentration (Cmax) of AU-007 | Day 1 thru EOT visit (28 days after last dose)
  The Cmax of AU-007 will be measured at different timepoints after AU-007 administration
Magnitude of PK changes in the blood after dosing determined by time of maximum concentration (Tmax) | Day 1 thru EOT visit (28 days after last dose)
  The Tmax of AU-007 will be measured at different timepoints after AU-007 administration
Magnitude of PK changes in the blood after dosing determined by Half-life (T1/2) of AU-007 | Day 1 thru EOT visit (28 days after last dose)
  The T1/2 of AU-007 will be measured at different timepoints after AU-007 administration
Magnitude of cytokine changes in the blood after dosing | Day 1 thru EOT visit (28 days after last dose)
Magnitude of immunogenicity after dosing with AU-007 alone or in combination with aldesleukin, AU-007 in combination with aldesleukin and avelumab or nivolumab | Day 1 thru EOT visit (28 days after last dose)
  Assessed by summarizing the number of patients who develop detectable anti-drug antibodies (ADAs) at different timepoints after AU-007 alone or in combination with aldesleukin, AU-007 in combination with aldesleukin and avelumab, or nivolumab
Evaluate the preliminary anti-tumor activity of AU-007 alone, in combination with aldesleukin, in combination with aldesleukin and avelumab, and AU-007 plus aldesleukin with nivolumab in patients with unresectable locally advanced or metastatic cancer | Day 1 thru EOT visit (28 days after last dose)
  Clinical anti-tumor activity will be evaluated using conventional Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and modified RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: James Vasselli, MD, Study Chair — Aulos Bioscience, Inc.
Locations (16):
- United States (9):
  - START Midwest, Grand Rapids, Michigan
  - Minnesota Oncology and Hematology PA, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Carolina Biooncology Institute, Huntersville, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology (Balcones) - SCRI, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - START South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (7):
  - Southside Cancer Care Centre, Miranda, New South Wales
  - Southern Oncology Clinical Research Unit, Bedford Park, South Australia
  - Monash Health, Clayton, Victoria
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Sunshine Hospital, Saint Albans, Victoria